CLINICAL TRIAL: NCT03890003
Title: An Early Feasibility Study to Evaluate the Predictive Low Glucose Suspend Functionality and Safety in an Automated Insulin Delivery System in Adult Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of an Automated Insulin Delivery System in Adult Participants With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17176; F3Z-MC-IORC (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- AID System Containing Insulin Lispro (Experimental): The automated insulin delivery (AID) system is comprised of a continuous subcutaneous insulin infusion (CSII) pump component with a PLGS algorithm, and a continuous glucose monitor (CGM) component.
  Interventions: Device: AID System; Drug: Insulin Lispro

INTERVENTIONS:
Device: AID System — AID system
  Other Names: LY8888AU
Drug: Insulin Lispro — Individualized doses of insulin lispro administered via the AID system to maintain glycemic control, except during procedures designed to induce hyperglycemia and hypoglycemia.
  Other Names: LY275585

SUMMARY:
The purpose of this early feasibility study is to assess the predictive low glucose suspend (PLGS) feature's safety, functionality and performance.

ELIGIBILITY:
Inclusion Criteria:

* Participants with T1DM for at least 2 years and who have used an insulin delivery system with any rapid-acting insulin analog for the preceding 6 months
* Have a body mass index of 18.5 to 37 kilogram per meter squared
* Have a hemoglobin A1c level ≥6.0% and ≤9.0%

Exclusion Criteria:

* Have known allergies or history of hypersensitivity to insulin lispro
* Have had an episode of severe hypoglycemia within the past 6 months
* Have had more than 1 episode of diabetic ketoacidosis in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) | In-Patient Period (2 Days)
  Number of AEs
Continuous Glucose Monitor (CGM) Measured Percentage of Time <70 mg/dL | In-Patient Period (2 Days)
  CGM measured percentage of time <70 milligrams per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinsker JE, Bartee A, Katz M, Lalonde A, Jones R, Dassau E, Wolpert H. Predictive Low-Glucose Suspend Necessitates Less Carbohydrate Supplementation to Rescue Hypoglycemia: Need to Revisit Current Hypoglycemia Treatment Guidelines. Diabetes Technol Ther. 2021 Jul;23(7):512-516. doi: 10.1089/dia.2020.0619. Epub 2021 Feb 18. PMID 33535013